CLINICAL TRIAL: NCT04544852
Title: Uncovering and Overcoming the Barriers of Colorectal Cancer Screening Amongst Spouses of Patients With Colorectal Cancer Through a Randomized Control Trial
Brief Title: Uncovering and Overcoming the Barriers of Colorectal Cancer Screening Amongst Spouses of Patients With Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, KER-KAN TAN, Assistant Professor Tan Ker Kan, National University Health System, Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: R-176-000-211-511
Record Dates: First submitted 2019-09-05; First posted 2020-09-10 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current practice (Placebo Comparator): "Intervention A" depicts current practices by informing the participants that FIT kits can be obtained from from the Singapore Cancer Society (SCS) or one of their collection point free of charge.
  Interventions: Behavioral: Current practice
- Targeted intervention programme (Active Comparator): "Intervention B" involves a targeted intervention programme tackling issues relating to a lack of education, inconvenience and cost would improve screening rates amongst the spouses.
  Interventions: Behavioral: Targeted intervention programme

INTERVENTIONS:
Behavioral: Current practice — "Intervention A" depicts current practices by informing the participants that FIT kits can be obtained from from the Singapore Cancer Society (SCS) or one of their collection point free of charge. Participants will be contacted at 3 months after enrollment to determine whether they have completed the FIT test.
  Arms: Current practice
Behavioral: Targeted intervention programme — The targeted intervention programme includes participants undergoing a structured educational program regarding colorectal cancer and the importance of screening in its prevention. The details will be explained to them using the pamphlet from MOH on Colorectal Cancer Screening. They will also be offered two FIT kits free of charge. Research team will educate participants on how to perform the FIT test. A detailed information guide on how to collect stool samples for FIT kit and how to return the completed FIT kit to the NUH Colorectal Centre will be given to them. Participants will be contacted at 3 months after enrollment to determine whether they have completed the FIT test.
  Arms: Targeted intervention programme

SUMMARY:
To determine amongst spouses of colorectal cancer patients:

1. Screening rates for Colorectal Cancer (CRC) amongst spouses of patients with CRC
2. Barriers to screening based on the Health Belief Model (HBM)
3. Mediators to behaviour change using the transtheoretical model of behavioural change
4. If tailored interventions addressing education, convenience and cost would improve screening rates amongst the spouses

DETAILED DESCRIPTION:
Stage 1: Randomization into Intervention versus Control

The eligible participants will be randomized into either "Intervention" or "Control" after the study team obtains participants' informed consent and before they begin doing the questionnaires. A randomisation list is generated using a computer procedure using block randomization. Based on the randomisation list, the assigned groups for each study participant's ID are written in a sealed opaque envelope. The envelope will be open at the point of randomisation to find out which group participant is randomised to.

The "Intervention" arm is aimed at specifically addressing gaps in terms of knowledge of colorectal cancer and the importance of screening, as well as targeting cost as well as convenience issues. Spouses who have been randomized into this arm will undergo a session with a trained research assistant who will highlight the following points:

1. What is colorectal cancer and what are its risk factors?
2. What is the spouse possibly at risk of developing colorectal cancer?
3. How can screening help to reduce the risk of colorectal cancer?
4. What are the screening modalities for CRC?
5. What are FIT kits?
6. How to use FIT kits?
7. Where to return the FIT kits once they have been used?

All participants who have undergone the counseling session will then be given 2 x FIT kits (as recommended in the guidelines) free of charge, and also advised to mail the FIT kits back to the colorectal clinic in a pre-paid envelope once it has been used. By performing the above targeted interventions, we would have tackled issues relating to education, cost and convenience.

The "Control" arm is the current practice in the community where these participants would be informed that the FIT kits can be obtained from the Singapore Cancer Society (SCS) free of charge if they fulfil the screening criteria as stipulated in the MOH guidelines. The participants will be advised on the various locations to collect these FIT kits.

The endpoint for the "intervention" and the "control" arms is whether the spouses returned the FIT kits within 3 months from date of consent.

Stage 2: Questionnaires

After obtaining informed consent, the spouse would be asked to fill in the baseline demographic form. After that, they will be asked if they have undergone any prior screening as recommended by the MOH screening guidelines as stipulated earlier. Following that, a quantitative questionnaire utilizing the validated Health Belief Model would be administered to study the potential barriers to screening which may be faced by the spouses. This questionnaire is based on the 5 domains of the Health Belief Model which include perceived susceptibility to acquiring CRC, perceived severity of the disease, perceived benefit of going for screening, perceived barriers to action and cues to action. The response options for questions on these domains are categorized into "disagree", "agree" and "unsure".

A second questionnaire based on the transtheoretical model would then be implemented next. We would determine their stage in the transtheoretical model based on their responses. The basic questionnaire was based on previous published data. This questionnaire will take approximately 5 minutes to complete.

Faecal Occult Blood Test or Colonoscopy:

Never heard: Has not heard of FOBT or colonoscopy. Precontemplation: Never had an FOBT or last FOBT was more than a year ago or last colonoscopy was more than 10 years ago and not thinking about having an FOBT or colonoscopy in the next 2 months.

Contemplation: Never had an FOBT or last FOBT was more than a year ago or last colonoscopy was more than 10 years ago but thinking about having an FOBT or colonoscopy in the next 2 months.

Action: FOBT was within the last year or colonoscopy was within the last year. Maintenance: Has undergone two or more FOBTs in the past 2 years or has undergone at least two or more colonoscopies and would continue to do so in concordance with the schedule

The same questionnaire would be repeated in 3 months and 6-12 months following the initial interview, with at least 3 months between each follow-up. This is in sync with the appointments that the patients themselves would be attending as part of their surveillance for their CRC. This is to document the changes in their responses to the various domains as the impact of the patients' cancers is less felt with time. The responses would guide the research team to determine if the peri-operative period remains the best time to advise the spouses to undergo screening or if we should delay it to a more appropriate and hence receptive period.

ELIGIBILITY:
Inclusion Criteria:

1. Has a partner who was diagnosed and treated for Colorectal Cancer
2. Either Singaporean or Permanent Resident;
3. Fulfilled the eligibility to undergo screening for colorectal cancer as stipulated by MOH.

Exclusion Criteria:

1. Pre-existing family history of FAP, HNPCC or inflammatory bowel disease in the family, as this would place the patient in the high risk group
2. Previous personal history of colorectal cancer or colorectal polyps
3. Underwent previous FOBT/FIT tests for CRC (this is an exclusion to participate in Stage 2-RCT only. Participants can still take part in Stage 1 and Stage 3 of the study if they fulfilled inclusion criteria 1-3, and did not meet any of the exclusion criteria 1-2)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-12-04 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants that completed the FIT test within three months post enrollment. | 3 months
  The research team would like to compare the percentage of FIT kit uptake rates amongst the two intervention arms. A positive outcome would be a higher percentage of FIT uptake seen in the targeted intervention arm.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Kent Ridge, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lau J, Choe L, Hui Juan Lee D, Khoo AM, Koh WL, Peh C, Ng A, Lim TZ, Lieske B, Lee KC, Chong CS, Seow CS, Keh CHL, Ng JY, Tan KK. Increasing Colorectal Screening Uptake in Spouses of Patients With Colorectal Cancer Using a Randomized Behavioral Trial. J Natl Compr Canc Netw. 2024 Jul 29;22(6):e247018. doi: 10.6004/jnccn.2024.7018. PMID 39074504